CLINICAL TRIAL: NCT04488601
Title: Participatory Evaluation (of) Aging (With) Rapamycin (for) Longevity Study (PEARL): A Prospective, Double-Blind, Placebo-Controlled Trial for Rapamycin in Healthy Individuals Assessing Safety and Efficacy in Reducing Aging Effects
Brief Title: Participatory Evaluation (of) Aging (With) Rapamycin (for) Longevity Study
Acronym: PEARL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AgelessRx (Industry)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ALRx001
Record Dates: First submitted 2020-07-13; First posted 2020-07-28 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2022-10

CONDITIONS: Aging
Keywords: rapamycin; aging; longevity; sirolimus; healthy aging; age-related conditions
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Intervention Model Description: Prospective, Double-Blind, Placebo-Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Rapamycin 5 (Experimental): Rapamycin 5 mg/week
  Interventions: Drug: Rapamycin
- Rapamycin 10 (Experimental): Rapamycin 10 mg/week
  Interventions: Drug: Rapamycin
- Placebo 1 (Placebo Comparator): Placebo once per week
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rapamycin — Rapamycin in 2 different dosage forms.
  Other Names: Sirolimus; Rapamune; Rapacan; Siromus; Raparen; Rapasim; Sirova
  Arms: Rapamycin 10; Rapamycin 5
Drug: Placebo — Placebo capsules
  Arms: Placebo 1

SUMMARY:
This is a randomized, placebo-controlled trial into the safety and efficacy in reducing clinical measures of aging in an older adult population.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled trial assessing the effects of low and high doses of intermittent Rapamycin on a weekly schedule. The researchers aim to establish a long-term safety profile, determine the long-term efficacy of Rapamycin in reducing clinical aging measures, and biochemical and physiological endpoints associated with declining health and aging in healthy older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-85
* Any sex
* Any ethnicity
* Interest in taking Rapamycin off-label
* Willing to undergo tests
* Relatively good health with only well-managed chronic diseases (hypertension, coronary artery disease, type II diabetes, etc.) clinically stable
* Adequate cognitive function to be able to give informed consent
* Technologically competent to complete web forms and perform video calls with the PI

Exclusion Criteria:

* Anemia - Hg < 9.0 g/dl, Leukopenia - white blood cells (WBC) < 3,500/mm3 , Neutropenia - absolute neutrophil count < 2,000/mm3 , or Platelet count - platelet count < 125,000/mm3
* Premenopausal females (due to menstruation-induced anemia, etc.)
* Patients scheduled to undergo major surgery in the next 12 months
* Patients undergoing or scheduled to undergo chemotherapy or any other treatment for malignancy
* Patients scheduled for immunosuppressant therapy for transplant
* Patients with impaired wound healing or history of a chronic open wound
* Untreated dyslipidemia with LDL-c > 190 and family history of dyslipidemia, Total cholesterol > 350 mg/dl, or triglycerides > 880 mg/dl.
* Impaired hepatic function, including elevated alkaline Phosphatase levels, aspartate aminotransferase (AST), alanine aminotransferase (ALT), Albumin, or T. Bili.
* HIV/AIDS, chronic Lyme, Babesia, Ehrlichiosis, Anaplasmosis, or other chronic infections that require ongoing treatment or monitoring
* Allergy to Rapamycin
* Any form of clinically relevant primary or secondary immune dysfunction or deficiency (e.g. X-linked agammaglobulinemia (XLA), common variable immunodeficiency (CVID))
* Chronic oral corticosteroid or immunosuppressive medication use (e.g. Enbrel, Humira, methotrexate).
* Fibromyalgia or Chronic Fatigue Syndrome/Myalgic Encephalomyelitis, Breast Implant Illness,
* Congestive heart failure: self-assessed functional status of heart failure New York Heart Association (NYHA) classification III or IV
* Impaired renal function, as defined as glomerular filtration rate (GFR) < 30
* Poorly controlled diabetes, as defined as HbA1c > 7%
* Type I Diabetes, or Insulin-dependent Type II diabetes
* Substance abuse disorder either untreated or if treated within the last 5 years
* PTSD, Bipolar disorder, Schizophrenia, or any other untreated or poorly controlled mental health or mood disorder, or history of hospitalization due to mental health condition
* Those who have taken metformin, rapamycin, or rapalogs in the past 6 months

  * (volunteers who were on metformin for aging can participate, provided they agree to stop taking metformin before and during the trial)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Changes in visceral fat as measured by dual-energy x-ray absorptiometry (DXA) scan | 6 month interim analysis of the data, 12 month safety profile will be established
  Visceral fat changes from baseline as determined by DXA scan.

SECONDARY OUTCOMES:
bone density | 6 month interim analysis of the data, 12 month safety profile will be established
  Changes in bone density from baseline as determined by DXA scan
lean body mass | 6 month interim analysis of the data, 12 month safety profile will be established
  Changes in lean body mass from baseline as determined by DXA scan
adverse events | 6 month interim analysis of the data, 12 month safety profile will be established
  Number of patients with adverse events using standard AE reporting (FDA regulations 21CFR314.80 and 1CFR213.32(s))
complete blood count (CBC) | 6 month interim analysis of the data, 12 month safety profile will be established
  changes in CBC from baseline
Change of blood electrolytes（serum potassium, sodium, chloride, and carbon dioxide in mmol/L）measured at baseline and after 6 and 12 months. | 6 month interim analysis of the data, 12 month safety profile will be established
  Difference in the change of blood electrolytes（serum potassium, sodium, chloride, and carbon dioxide in mmol/L) compared with the baseline at 6 and 12 months between the intervention and control group is to be analyzed.
Change of liver function as measured by serum globulin in g/dL, measured at baseline and after 6 and 12 months. | 6 month interim analysis of the data, 12 month safety profile will be established
  Difference in the change of liver function as measured by serum globulin in g/dL compared with the baseline at 6 and 12 months between the intervention and control group is to be analyzed.
Change of liver function as measured by serum bilirubin in mg/dL, measured at baseline and after 6 and 12 months. | 6 month interim analysis of the data, 12 month safety profile will be established
  Difference in the change of liver function as measured by serum bilirubin in mg/dL compared with the baseline at 6 and 12 months between the intervention and control group is to be analyzed.
Change of liver function as measured by serum alkaline phosphatase, AST, and ALT in IU/L, measured at baseline and after 6 and 12 months. | 6 month interim analysis of the data, 12 month safety profile will be established
  Difference in the change of liver function as measured by serum alkaline phosphatase, AST, and ALT in IU/L compared with the baseline at 6 and 12 months between the intervention and control group is to be analyzed.
Change of renal function as measured by serum albumin in g/dL, measured at baseline and after 6 and 12 months. | 6 month interim analysis of the data, 12 month safety profile will be established
  Difference in the change of renal function as measured by serum albumin in g/dL compared with the baseline at 6 and 12 months between the intervention and control group is to be analyzed.
Change of renal function as measured by serum creatinine and uric acid in mg/dL, measured at baseline and after 6 and 12 months. | 6 month interim analysis of the data, 12 month safety profile will be established
  Difference in the change of renal function as measured by serum creatinine and uric acid in mg/dL compared with the baseline at 6 and 12 months between the intervention and control group is to be analyzed.
Change in lipids (serum total cholesterol, triglycerides, HDL, and LDL cholesterol in mg/dL) measured at baseline and after 6 and 12 months. | 6 month interim analysis of the data, 12 month safety profile will be established
  Difference in the change of lipids（serum total cholesterol, triglycerides, HDL and LDL cholesterol in mg/dL) compared with the baseline at 6 and 12 months between the intervention and control group is to be analyzed.
Change in fasting serum glucose in mg/dL, measured at baseline and after 6 and 12 months. | 6 month interim analysis of the data, 12 month safety profile will be established
  Difference in the change of fasting serum glucose in mg/dL compared with baseline at 6 and 12 months between the intervention and control group is to be analyzed.
Change in insulin in uIU/mL, measured at baseline and after 6 and 12 months. | 6 month interim analysis of the data, 12 month safety profile will be established
  Difference in the change of fasting serum insulin in uIU/mL compared with baseline at 6 and 12 months between the intervention and control group is to be analyzed.
Change in fasting serum IGF-1 in ng/mL, measured at baseline and after 6 and 12 months. | 6 month interim analysis of the data, 12 month safety profile will be established
  Difference in the change of fasting serum IGF-1 in ng/mL compared with baseline at 6 and 12 months between the intervention and control group is to be analyzed.
Change in serum Hemoglobin A1c in % of total hemoglobin, measured at baseline and after 6 and 12 months. | 6 month interim analysis of the data, 12 month safety profile will be established
  Difference in the change of serum Hemoglobin A1c in % of total hemoglobin compared with baseline at 6 and 12 months between the intervention and control group is to be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: James Watson, MD, Principal Investigator — University of California, Los Angeles; Sajad Zalzala, MD, Study Director — AgelessRx
Locations (1):
- AgelessRx, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: as soon as available
Access Criteria: Institutional review board (IRB) approval or at the discretion of PI/sponsor